CLINICAL TRIAL: NCT03385018
Title: Multicenter Randomized Controlled Trial for Application of Laparoscopic Total Gastrectomy With Lymph Node Dissection for Gastric Cancer (KLASS-06)
Brief Title: Trial for Application of Laparoscopic Total Gastrectomy With Lymph Node Dissection for Gastric Cancer (KLASS-06)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2017-0940
Record Dates: First submitted 2017-12-20; First posted 2017-12-28 (Actual); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Intervention Model Description: 2-arm randomized controlled study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laparoscopic group (Experimental): Arm Description: Laparoscopic radical total gastrectomy with D2 (or D2-#10) lymph node dissection
  Interventions: Procedure: Radical total gastrectomy with D2 (D2 - #10) lymph node dissection by laparoscopic approach
- Open group (Active Comparator): Open radical total gastrectomy with D2 (or D2-#10) lymph node dissection
  Interventions: Procedure: Radical total gastrectomy with D2 (D2 - #10) lymph node dissection by open conventional approach

INTERVENTIONS:
Procedure: Radical total gastrectomy with D2 (D2 - #10) lymph node dissection by laparoscopic approach — * Total gastrectomy with D2(D2-10) lymph node dissection by laparoscopic approach
  * The number of trocars is 6 or less
  * Roux-en-Y esophagojejunostomy with any stapling method
  * Enough(negative) margin from tumor
  * LN station #1, 2, 3, 4d, 4sb, 5, 6, 7, 8a, 9, (10), 11p, 11d, 12a should be examined
  * Washing cytology
  * Frozen biopsy for surgical margin at surgeons discretion
  * Complete omentectomy for grossly serosa-involved tumor
  * Combined organ resection only in cholecystectomy and splenectomy
  * Indwelling nasogastric tube and drainage catheter at surgeons discretion
  * D2 lymphadenectomy should be performed : dissection of LN stations No.4d, 4sb, 4sa, 2, 10 (splenic hilar LN can be left according to the clinical stage), 6, 5, 12a, 8a, 9, 7, 1, 3, 11p, 11d with prevention of pancreatic injury during suprapancreatic dissection
  Arms: Laparoscopic group
Procedure: Radical total gastrectomy with D2 (D2 - #10) lymph node dissection by open conventional approach — * Total gastrectomy with D2(D2-10) lymph node dissection by open conventional approach
  * Roux-en-Y esophagojejunostomy with any stapling method
  * Enough(negative) margin from tumor
  * LN station #1, 2, 3, 4d, 4sb, 5, 6, 7, 8a, 9, (10), 11p, 11d, 12a should be examined
  * Washing cytology
  * Frozen biopsy for surgical margin at surgeons discretion
  * Complete omentectomy for grossly serosa-involved tumor
  * Indwelling nasogastric tube and drainage catheter at surgeons discretion
  * D2 lymphadenectomy should be performed : dissection of LN stations No.4d, 4sb, 4sa, 2, 10 (splenic hilar LN can be left according to the clinical stage), 6, 5, 12a, 8a, 9, 7, 1, 3, 11p, 11d with prevention of pancreatic injury during suprapancreatic dissection
  Arms: Open group

SUMMARY:
Although Laparoscopic gastrectomy for both early and locally advanced gastric cancer has gained popularity, the use of laparoscopic total gastrectomy for proximal advanced gastric cancer is still limited to some experienced surgeons, because of its technical difficulties in D2 lymph node dissection and anastomoses.

Some retrospective and cohort studies regarding laparoscopic total gastrectomy with lymph node dissection suggested the likelihood of application of laparoscopic surgery for proximal gastric cancer. However, there has been no randomized clinical trial comparing results of laparoscopic total gastrectomy with D2 lymph node dissection with open conventional surgery.

Therefore, we aimed to verify the efficacy of laparoscopic total gastrectomy with D2(D2-10) lymph node dissection, technical and oncologic safety compared with open surgery via multicenter randomized clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are over 20 and below 80 years old
* Patients who have performance status of ECOG 0 or 1
* Patients with American Society of Anesthesiology score of class I to III
* Patients who are diagnosed with gastric adenocarcinoma not involving Z-line by endoscopy with biopsy
* Patients with tumors which can be curatively resected by total gastrectomy with lymph node dissection based on preoperative study
* Patients who have primary gastric carcinoma invaded into over muscle propria, and not into adjacent organ in preoperative studies (cT2 ~ cT4a)
* Patients who have no metastasis to lymph nodes or limited metastasis to perigastric lymph node metastasis in preoperative studies (cN0 ~ cN2)
* Patients who agree with participating in the clinical study with informed consents
* Patients who can be followed for at least 3 years after study enrollment

Exclusion Criteria:

* Patients who have possibility of distant metastasis in preoperative studies
* Patients who have history of gastric resection with any cause
* Patients who have complications (bleeding or obstruction) of gastric cancer
* Patients who are treated by chemo(radio)therapy or endoscopic submucosal dissection for gastric cancer
* Patients who are diagnosed and treated with other malignancies within 5 years
* Vulnerable patients
* Patients who participating or participated in other clinical trial within 6 months

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 772 (Estimated)
Dates: Start 2018-04-05 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
3 year relapse-free survival | 3 years after surgery
  Non-inferiority of 3 year relapse-free survival rate after laparoscopic radical total gastrectomy and lymphadenectomy for locally advanced gastric cancer comparing with open conventional surgery.
  The "event" of relapse-free survival is defined as "recurrence" after 4 weeks of operation.
  The "censoring" is defined as non-traceable patient who cannot be confirmed with recurrence or patient who are alive without recurrence until follow-up.
  The "relapse-free survival time" is defined as the time from surgery to "event" or "censoring".

SECONDARY OUTCOMES:
3 year overall survival rate | 3 years after surgery
5 year relapse-free and overall survival | 5 years after surgery
Morbidity (early period) | from Operation day until POD 21
Morbidity (late period) | from POD (Post-Operative Day) 22 until 5 years after surgery
Mortality | at POD 30
  death with any cause
Mortality | at POD 90
  death with any cause
Quality of life(EORTC QLQ-C30) | at POD 21
  Quality of life measured by EORTC QLQ-C30(Version 3) The questionnaire was designed to measure cancer patients' physical, psychological and social functions. The questionnaire is composed of 5 multiitem scales (physical, role, social, emotional and cognitive functioning) and 9 single items (pain, fatigue, financial impact, appetite loss, nausea/vomiting, diarrhea, constipation, sleep disturbance and quality of life).
Quality of life(EORTC QLC STO22) | at POD 21
  Quality of life measured by EORTC QLC STO22. The EORTC QLQ-STO 22 module contains 22 items in a similar layout and response format to the EORTC QLQ-C30. The hypothesised scale structure of the module consists of five scales (dysphagia, eating restrictions, pain, reflux and anxiety) and three single items (dry mouth, body image and hair loss).
Quality of life(EORTC QLQ-C30) | 3 months after surgery
  Quality of life measured by EORTC QLQ-C30(Version 3)
Quality of life(EORTC QLC STO22) | 3 months after surgery
  Quality of life measured by EORTC QLC STO22. The EORTC QLQ-STO 22 module contains 22 items in a similar layout and response format to the EORTC QLQ-C30. The hypothesised scale structure of the module consists of five scales (dysphagia, eating restrictions, pain, reflux and anxiety) and three single items (dry mouth, body image and hair loss).
Quality of life(EORTC QLQ-C30) | 12 months after surgery
  Quality of life measured by EORTC QLQ-C30(Version 3)
Quality of life(EORTC QLC STO22) | 12 months after surgery
  Quality of life measured by EORTC QLC STO22. The EORTC QLQ-STO 22 module contains 22 items in a similar layout and response format to the EORTC QLQ-C30. The hypothesised scale structure of the module consists of five scales (dysphagia, eating restrictions, pain, reflux and anxiety) and three single items (dry mouth, body image and hair loss).

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Surgery, Yonsei University College of Medicine, Seoul, Korea, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No